CLINICAL TRIAL: NCT03593473
Title: The Psychobiology of Resilience in Mother-child Pairs: Inhaled Oxytocin and HPA Axis Reactivity
Brief Title: Inhaled Oxytocin and HPA Axis Reactivity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 12-2061; R01HD093901-01A1 (NIH)
Record Dates: First submitted 2018-06-05; First posted 2018-07-20 (Actual); Results first posted 2024-05-24 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2024-04

CONDITIONS: Depression, Postpartum; Anxiety Disorders; Stress, Psychological
Keywords: Oxytocin; Hypothalamic-pituitary-adrenal axis (HPA)
MeSH Terms: conditions — Depression, Postpartum; Anxiety Disorders; Stress, Psychological | interventions — Oxytocin

STUDY DESIGN:
Intervention Model Description: Non-pregnant women will be randomized to either 24 IU of nasal OT or placebo. The Investigational Drug Service will use a random number generator to prepare a randomization table.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will receive a nasal insufflation bottle of oxytocin intranasal spray or placebo intranasal spray manufactured to mimic oxytocin nasal spray.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Intranasal Oxytocin (Experimental): Participants block randomized to Oxytocin intranasal spray by risk status at enrollment in the Mood, Mother and Infant (MMI) study and as verified by structured clinical diagnostic interview (no history of depression or anxiety, past depression or anxiety, current depression or anxiety).
  Interventions: Drug: Intranasal Oxytocin
- Placebo (Placebo Comparator): Participants block randomized to placebo Intranasal spray with all equivalent ingredients except oxytocin. Blocks will be stratified by risk status at enrollment in the Mood, Mother and Infant (MMI) study and as verified by structured clinical diagnostic interview (no history of depression or anxiety, past depression or anxiety, current depression or anxiety).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Intranasal Oxytocin — Six intranasal sprays of oxytocin. Each insufflation delivers 4 IUs of oxytocin for a total oxytocin dosage of 24 IUs.
  Other Names: Syntocinon
  Arms: Intranasal Oxytocin
Drug: Placebo — Six intranasal sprays of placebo manufactured to mimic oxytocin nasal spray containing all equivalent ingredients except oxytocin.
  Other Names: Inactive
  Arms: Placebo

SUMMARY:
Mothers who were enrolled in the Mood, Mother and Infant study will be eligible to participate in the 6-year follow-up maternal visit. At the time of this visit, mothers will be randomized to a single 24 IU dose of nasal oxytocin or placebo. Following administration of the study drug, women will participate in the Trier Social Stress Test (TSST), and blood samples will be collected to quantify HPA axis reactivity.

DETAILED DESCRIPTION:
The Mood, Mother and Infant Study is a prospective observational cohort study that began enrollment in May of 2013. Women were recruited in the 3rd trimester of pregnancy and followed prospectively through 12 months postpartum. Mother-infant pairs who completed the 12-month visit will be invited to participate in the current Psychobiology of Resilience in Maternal-Child Pairs follow-up study. The trial described here is a randomized controlled trial embedded within the Psychobiology of Resilience study.

Non-pregnant women will be randomized to either 24 IU of nasal oxytocin (OT) or placebo. The Investigational Drug Service (IDS) will use a random number generator to prepare a randomization table. Participants will be block randomized by risk status at enrollment in the Mood, Mother and Infant (MMI) study, as verified by structured clinical diagnostic interview (No history of depression or anxiety, Past depression or anxiety, current depression or anxiety). Both participants and study personnel will be blinded to allocation group. At the end of the protocol, participants will be asked which condition they believed they were in ('oxytocin,' 'control,' 'not sure') to ascertain success of blinding. Forty minutes after treatment, women will undergo the Trier Social Stress Test (TSST), comprised of a speech task and a math task; the TSST reliably induces large and consistent HPA and cardiovascular responses. The TSST is administered as follows: Pre-Task Instructions: (5 minutes) Subjects will be introduced to 3 people (the 'selection committee') and asked to assume the role of a job applicant. Anticipation Period: The subject prepares her speech for 3 minutes in the presence of the committee. Speech: The committee asks the subject to deliver her talk for 5 minutes while being video and audio-recorded. If the subject finishes early, the committee responds with prepared questions to ensure that she speaks for the entire 5 minutes. These questions are designed to be non-harassing but to create a feeling of lack of predictability/controllability (e.g., "Do you have any enemies?") Serial Subtraction (PASST): The committee will ask the subject to subtract the number 7 from 2000 as quickly and accurately as possible for 5 minutes. For each mistake, the committee says "Stop -- mistake -- start over at 2000." Stress Recovery: The subject sits quietly alone for 20 minutes.

Blood will be collected at baseline, during the speech and math tasks, and at 10 and 20 minutes of recovery, as HPA-axis responses are reliably found 10-30 minutes following the TSST. Evidence regarding optimal timing of stress testing is conflicting. Visits will be scheduled for 1 pm to increase likelihood of detecting a stress response unopposed by the circadian influence, based on the experience of investigators in our laboratory and published studies of postpartum women. These investigators have found menstrual cycle phase does not affect TSST results; therefore, the date of last menstrual period and hormone use will be recorded, but visits will not be scheduled based on cycle phase.

ELIGIBILITY:
This study will follow-up the existing Mood, Mother and Infant (MMI) prospective longitudinal cohort (R01HD073220), comprised of 222 mother-infant dyads who were recruited between May 2013 and April 2017 and completed the 12-month MMI visit. In the MMI study, 222 mothers ages 18-45 and their infants were enrolled. Participants were recruited from community clinics in the third trimester of pregnancy and continued to participate in the study through 12 months postpartum. At the 12-month visit, mothers were invited to continue to be followed via online surveys at 6-month intervals; more than 80% of women who have completed the MMI study to date have continued to participate. Enrolled participants in the MMI study met the following inclusion and exclusion criteria:

Inclusion Criteria:

1. Singleton pregnancy;
2. Intention to breastfeed (due to the centrality of breastfeeding to the oxytocin assessment);
3. Intention to remain within 40 miles of the University of North Carolina - Chapel Hill through infant's first birthday;
4. Ability to communicate in English.

Exclusion Criteria:

1. Maternal diagnosis of Axis I disorders other than unipolar depression or anxiety disorders. Women with a history of bipolar disorder were excluded, given their increased risk of postpartum psychosis.
2. Active substance abuse at enrollment in the 3rd trimester of pregnancy (Tobacco, alcohol, illicit substances);
3. Major congenital anomaly;
4. Chronic medication/medical condition contraindicated for breastfeeding;
5. Current use of tricyclic antidepressants, which alter cortisol and heart rate variability.

At enrollment, all participants underwent a Structured Clinical Interview Non-Patient version (SCID-NP).

Inclusion Criteria for Inhaled Oxytocin and HPA Axis Reactivity, a substudy of the Psychobiology of Resilience in Mother-Child Pairs follow-up study: 1) Participated in the MMI study 2) Both mother and child willing and able to participate in the 6-year follow-up visits 3) Not pregnant, verified by urine pregnancy test on day of study visit.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2019-02-07 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison M Stuebe, MD, MSc, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina School of Medicine, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared according to the most recent NIH guidelines.
Supporting Information: Study Protocol
Time Frame: Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB) and executes a data use/sharing agreement with the University of North Carolina (UNC).
Access Criteria: Individual level data sharing will be subject to local IRB approval, individual written informed consents, and national law
URL: http://mmi.web.unc.edu

REFERENCES:
- [Derived] Mills-Koonce WR, Grewen K, O'Shea NG, Pearson B, Strange CG, Meltzer-Brody SE, Guintivano JD, Stuebe AM. The Mood, Mother and Child Study: Protocol for a Prospective Longitudinal Study and Randomized Controlled Trial. JMIR Res Protoc. 2023 Oct 26;12:e51132. doi: 10.2196/51132. PMID 37883133
- See also: Mood, mother and infant study web site — http://mmi.web.unc.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intranasal Oxytocin | Placebo
Started | 53 | 56
Randomized | 53 | 56
Received Intervention | 51 | 54
Completed | 51 | 54
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intranasal Oxytocin | Placebo | Total
Number analyzed (Participants) | 51 | 54 | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.63 (4.38) | 38.26 (3.98) | 37.95 (4.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 54 | 105
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 10
  Not Hispanic or Latino | 46 | 49 | 95
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 8 | 3 | 11
  White | 40 | 44 | 84
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 51 | 54 | 105

OUTCOME MEASURES:

1. Primary Outcome: Mean Cortisol (CRT) During Trier Social Stress Test (TSST)
Description: The study drug will be administered 40 minutes before the TSST. Serum cortisol will be measured via peripheral IV 40 (-40) and 20 (-20) minutes before the TSST, at the start of the TSST (0 minutes), and at minutes 10 (during the speech task), 15 (during the math task), 28, 38, and 48 (during recovery).
Time Frame: -40 minutes, -20 minutes, 0 minutes, +10 minutes, +15 minutes, +28 minutes, +38 minutes, +48 minutes
Population: Samples were collected by IV. In some participants, an IV was not able to be placed and samples could not be collected. In some participants, an IV was successfully placed, but the IV infiltrated before the end of the observation period and not all timepoints were collected. One participant had a vasovagal episode when the IV was placed and samples were not collected. All collected data are reported herein.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Intranasal Oxytocin | Placebo
Number analyzed (Participants) | 42 | 47
pg/mL
  -40 minutes | 19.17 (13.46) | 16.87 (10.84)
  -20 minutes: number analyzed (Participants) | 41 | 45
  -20 minutes | 15.71 (10.16) | 13.89 (9.68)
  0 minutes: number analyzed (Participants) | 41 | 43
  0 minutes | 14.06 (10.41) | 13.03 (8.99)
  +10 minutes: number analyzed (Participants) | 41 | 42
  +10 minutes | 14.39 (10.55) | 13.60 (9.45)
  +15 minutes: number analyzed (Participants) | 40 | 42
  +15 minutes | 15.27 (12.56) | 15.64 (10.16)
  +28 minutes: number analyzed (Participants) | 38 | 39
  +28 minutes | 16.78 (13.63) | 16.29 (9.44)
  +38 minutes: number analyzed (Participants) | 38 | 36
  +38 minutes | 14.50 (12.02) | 15.40 (9.66)
  +48 minutes: number analyzed (Participants) | 35 | 37
  +48 minutes | 13.16 (9.35) | 14.41 (9.02)
Statistical Analysis 1: Comparison: Intranasal Oxytocin vs Placebo; T-test comparing mean cortisol by study arm at -40 minutes; Test type: Superiority; p = 0.37, t-test, 2 sided
Statistical Analysis 2: Comparison: Intranasal Oxytocin vs Placebo; T-test comparing mean cortisol by study arm at -20 minutes; Test type: Superiority; p = 0.40, t-test, 2 sided
Statistical Analysis 3: Comparison: Intranasal Oxytocin vs Placebo; T-test comparing mean cortisol by study arm at 0 minutes; Test type: Superiority; p = 0.63, t-test, 2 sided
Statistical Analysis 4: Comparison: Intranasal Oxytocin vs Placebo; T-test comparing mean cortisol by study arm at 10 minutes; Test type: Superiority; p = 0.72, t-test, 2 sided
Statistical Analysis 5: Comparison: Intranasal Oxytocin vs Placebo; T-test comparing mean cortisol by study arm at 15 minutes; Test type: Superiority; p = 0.88, t-test, 2 sided
Statistical Analysis 6: Comparison: Intranasal Oxytocin vs Placebo; T-test comparing mean cortisol by study arm at 28 minutes; Test type: Superiority; p = 0.85, t-test, 2 sided
Statistical Analysis 7: Comparison: Intranasal Oxytocin vs Placebo; T-test comparing mean cortisol by study arm at 38 minutes; Test type: Superiority; p = 0.72, t-test, 2 sided
Statistical Analysis 8: Comparison: Intranasal Oxytocin vs Placebo; T-test comparing mean cortisol by study arm at 48 minutes; Test type: Superiority; p = 0.57, t-test, 2 sided
Statistical Analysis 9: Comparison: Intranasal Oxytocin vs Placebo; A mixed effects model with random intercept and slope was used to model cortisol as the outcome variable with time, study arm, and an interaction between time and study arm as the exposure variables. Times are restricted to times 0, +10, +15, and +28, which reflect the measures taken during the Trier Social Stress Test. The p-value presented below is for the interaction term between time and study arm; Test type: Superiority; p = 0.96, Mixed Models Analysis

2. Secondary Outcome: Mean Adrenocorticotropic Hormone (ACTH ) During TSST
Description: The study drug will be administered 40 minutes before the TSST. Adrenocorticotropic hormone will be measured via peripheral IV 40 (-40) and 20 (-20) minutes before the TSST, at the start of the TSST (0 minutes), and at minutes 10 (during the speech task), 15 (during the math task), 28, 38, and 48 (during recovery).
Time Frame: -40 minutes, -20 minutes, 0 minutes, +10 minutes, +15 minutes, +28 minutes, +38 minutes, +48 minutes
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Intranasal Oxytocin | Placebo
Number analyzed (Participants) | 42 | 47
pg/mL
  -40 minutes | 79.96 (64.89) | 86.77 (103.00)
  -20 minutes: number analyzed (Participants) | 40 | 45
  -20 minutes | 85.73 (68.28) | 87.61 (92.74)
  0 minutes: number analyzed (Participants) | 41 | 43
  0 minutes | 84.31 (54.49) | 86.10 (93.42)
  +10 minutes: number analyzed (Participants) | 41 | 43
  +10 minutes | 80.31 (59.49) | 94.00 (86.89)
  +15 minutes: number analyzed (Participants) | 38 | 43
  +15 minutes | 93.46 (59.92) | 94.21 (104.00)
  +28 minutes: number analyzed (Participants) | 37 | 40
  +28 minutes | 84.02 (64.26) | 77.48 (87.08)
  +38 minutes: number analyzed (Participants) | 38 | 37
  +38 minutes | 79.38 (63.01) | 84.01 (81.48)
  +48 minutes: number analyzed (Participants) | 35 | 37
  +48 minutes | 77.27 (63.69) | 85.30 (74.79)
Statistical Analysis 1: Comparison: Intranasal Oxytocin vs Placebo; T-test comparing mean ACTH by study arm at -40 minutes; Test type: Superiority; p = 0.71, t-test, 2 sided
Statistical Analysis 2: Comparison: Intranasal Oxytocin vs Placebo; T-test comparing mean ACTH by study arm at -20 minutes; Test type: Superiority; p = 0.92, t-test, 2 sided
Statistical Analysis 3: Comparison: Intranasal Oxytocin vs Placebo; T-test comparing mean ACTH by study arm at 0 minutes; Test type: Superiority; p = 0.92, t-test, 2 sided
Statistical Analysis 4: Comparison: Intranasal Oxytocin vs Placebo; T-test comparing mean ACTH by study arm at 10 minutes; Test type: Superiority; p = 0.40, t-test, 2 sided
Statistical Analysis 5: Comparison: Intranasal Oxytocin vs Placebo; T-test comparing mean ACTH by study arm at 15 minutes; Test type: Superiority; p = 0.97, t-test, 2 sided
Statistical Analysis 6: Comparison: Intranasal Oxytocin vs Placebo; T-test comparing mean ACTH by study arm at 28 minutes; Test type: Superiority; p = 0.71, t-test, 2 sided
Statistical Analysis 7: Comparison: Intranasal Oxytocin vs Placebo; T-test comparing mean ACTH by study arm at 38 minutes; Test type: Superiority; p = 0.78, t-test, 2 sided
Statistical Analysis 8: Comparison: Intranasal Oxytocin vs Placebo; T-test comparing mean ACTH by study arm at 48 minutes; Test type: Superiority; p = 0.63, t-test, 2 sided
Statistical Analysis 9: Comparison: Intranasal Oxytocin vs Placebo; A mixed effects model with random intercept and slope was used to model cortisol as the outcome variable with time, study arm, and an interaction between time and study arm as the exposure variables. This is the p-value for the interaction term between time and study arm; Test type: Superiority; p = 0.11, Mixed Models Analysis

3. Secondary Outcome: Lagged Association Between ACTH and CRT During the TSST
Description: Correlations will be quantified between ACTH at time j and CRT at time j+1 to test the extent to which CRT response is blunted by exogenous oxytocin (OT).
Time Frame: ACTH at -40 minutes, -20 minutes, 0 minutes, +10 minutes, +15 minutes, +28 minutes, +38 minutes and Cortisol at -20 minutes, 0 minutes, +10 minutes, +15 minutes, +28 minutes, +38 minutes, +48 minutes
Population: as for outcome 1
Measure: Number; unit: Correlation coefficient
Arm/Group | Intranasal Oxytocin | Placebo
Number analyzed (Participants) | 41 | 44
Correlation coefficient
  ACTH at -40 minutes with Cortisol at -20 minutes | 0.07 | 0.44
  ACTH at -20 minutes with 0 minutes: number analyzed (Participants) | 40 | 42
  ACTH at -20 minutes with 0 minutes | 0.04 | 0.31
  ACTH at 0 minutes with Cortisol at +10 minutes: number analyzed (Participants) | 41 | 41
  ACTH at 0 minutes with Cortisol at +10 minutes | 0.16 | 0.46
  ACTH at +10 minutes with Cortisol at +15 minutes: number analyzed (Participants) | 40 | 42
  ACTH at +10 minutes with Cortisol at +15 minutes | 0.01 | 0.34
  ACTH at +15 minutes with Cortisol at +28 minutes: number analyzed (Participants) | 36 | 39
  ACTH at +15 minutes with Cortisol at +28 minutes | -0.04 | 0.40
  ACTH at +28 minutes with Cortisol at +38 minutes: number analyzed (Participants) | 37 | 36
  ACTH at +28 minutes with Cortisol at +38 minutes | 0.10 | 0.47
  ACTH at +38 minutes with Cortisol at +48 minutes: number analyzed (Participants) | 35 | 36
  ACTH at +38 minutes with Cortisol at +48 minutes | 0.29 | 0.26
Statistical Analysis 1: Comparison: Intranasal Oxytocin vs Placebo; Fisher's Z test for correlation between ACTH at -40 minutes and Cortisol at -20 minutes; Test type: Superiority; p = 0.07, Fisher's Z test
Statistical Analysis 2: Comparison: Intranasal Oxytocin vs Placebo; Fisher's Z test for correlation between ACTH at -20 minutes and Cortisol at 0 minutes; Test type: Superiority; p = 0.22, Fisher's Z test
Statistical Analysis 3: Comparison: Intranasal Oxytocin vs Placebo; Fisher's Z test for correlation between ACTH at 0 minutes and Cortisol at +10 minutes; Test type: Superiority; p = 0.14, Fisher's Z test
Statistical Analysis 4: Comparison: Intranasal Oxytocin vs Placebo; Fisher's Z test for correlation between ACTH at +10 minutes and Cortisol at +15 minutes; Test type: Superiority; p = 0.14, Fisher's Z test
Statistical Analysis 5: Comparison: Intranasal Oxytocin vs Placebo; Fisher's Z test for correlation between ACTH at +15 minutes and Cortisol at +28 minutes; Test type: Superiority; p = 0.05, Fisher's Z test
Statistical Analysis 6: Comparison: Intranasal Oxytocin vs Placebo; Fisher's Z test for correlation between ACTH at +28 minutes and Cortisol at +38 minutes; Test type: Superiority; p = 0.10, Fisher's Z test
Statistical Analysis 7: Comparison: Intranasal Oxytocin vs Placebo; Fisher's Z test for correlation between ACTH at +38 minutes and Cortisol at +48 minutes; Test type: Superiority; p = 0.90, Fisher's Z test
Statistical Analysis 8: Comparison: Intranasal Oxytocin vs Placebo; A mixed effects model with random intercept and slope was used to model cortisol at time j+1 as the outcome with ACTH at time j, study arm, and an interaction term between ACTH at time j and study arm as the exposure variables. The p-value presented below is for the interaction term between ACTH at time j and study arm; Test type: Superiority; p = 0.21, Mixed Models Analysis

4. Secondary Outcome: Changes in High Frequency Respiratory Sinus Arrhythmia Power, an Index of Parasympathetic Activity, During the TSST
Description: Recording of autonomic activity beginning prior to study drug administration (-40 minutes) until the end of recovery from the TSST (+38 minutes). Mobile Impedance Cardiographs (MindWare Tech Ltd, Gahanna, OH) was used to measure cardiac rate and interbeat interval (IBI). MindWare Heart Rate Variability (HRV) software was used to derive respiration and to calculate high frequency respiratory sinus arrhythmia power from the IBI series as an index of parasympathetic activity. Results are reported as difference from the mean of high frequency respiratory sinus arrhythmia power measured in the first ten minutes of the study visit, prior to administration of OT or placebo.
Time Frame: Minutes -40 to -35, -35 to -30, -30 to -25, -25 to -20, -20 to -15, -15 to -10, -10 to -5, -5 to 0, 5 to 8, 8 to 13, 13 to 18, 18 to 23, 23 to 28, 28 to 33, 33 to 38, 38 to 43, 43 to 48
Population: For two participants in each arm, cardiograph recording was unsuccessful. For some time periods for some participants, data quality or quantity (in terms of lacking sufficient numbers of epochs within a period) was insufficient for analysis. All valid, analyzable data are reported herein.
Measure: Mean (Standard Deviation); unit: ms squared
Arm/Group | Intranasal Oxytocin | Placebo
Number analyzed (Participants) | 49 | 52
ms squared
  -40 to -35 | 9.4867 (367.6) | 25.2298 (426.2)
  -35 to -30 | -54.8211 (341) | -76.7692 (476.9)
  -30 to -25 | 25.9791 (520.3) | -34.2107 (513.2)
  -25 to -20: number analyzed (Participants) | 49 | 49
  -25 to -20 | 8.1879 (412.4) | -85.2953 (494)
  -20 to -15: number analyzed (Participants) | 49 | 50
  -20 to -15 | 29.8191 (355.4) | -34.1119 (427.6)
  -15 to -10: number analyzed (Participants) | 49 | 50
  -15 to -10 | -65.0835 (303.9) | -50.8918 (363)
  -10 to -5: number analyzed (Participants) | 47 | 50
  -10 to -5 | -40.6283 (291) | -65.8414 (487.4)
  -5 to 0: number analyzed (Participants) | 47 | 48
  -5 to 0 | -66.7889 (365.5) | -0.2369 (440.3)
  5 to 8: number analyzed (Participants) | 49 | 48
  5 to 8 | -213.8 (577.3) | -60.7299 (424.1)
  8 to 13: number analyzed (Participants) | 49 | 48
  8 to 13 | -142.7 (729.6) | -93.6755 (585.2)
  13 to 18: number analyzed (Participants) | 49 | 49
  13 to 18 | -166 (702.4) | 45.2548 (701.9)
  18 to 23: number analyzed (Participants) | 47 | 48
  18 to 23 | -54.7814 (538.4) | 140.5 (416)
  23 to 28: number analyzed (Participants) | 47 | 47
  23 to 28 | -55.4212 (376.5) | 90.0612 (574.9)
  28 to 33: number analyzed (Participants) | 47 | 47
  28 to 33 | -2.1457 (484.3) | 78.347 (480)
  33 to 38: number analyzed (Participants) | 46 | 47
  33 to 38 | 10.4342 (551.7) | 94.173 (439.2)
  38 to 43: number analyzed (Participants) | 47 | 45
  38 to 43 | -31.2704 (497) | 74.8732 (390.8)
  43 to 48: number analyzed (Participants) | 47 | 44
  43 to 48 | -66.8297 (498.9) | 82.3593 (289.3)
Statistical Analysis 1: Comparison: Intranasal Oxytocin vs Placebo; High frequency heart rate variability at minutes -40 to -35; Test type: Superiority; p = 0.8441, t-test, 2 sided
Statistical Analysis 2: Comparison: Intranasal Oxytocin vs Placebo; High frequency heart rate variability at minutes -35 to -30; Test type: Superiority; p = 0.7919, t-test, 2 sided
Statistical Analysis 3: Comparison: Intranasal Oxytocin vs Placebo; High frequency heart rate variability at minutes -30 to -25; Test type: Superiority; p = 0.5639, t-test, 2 sided
Statistical Analysis 4: Comparison: Intranasal Oxytocin vs Placebo; High frequency heart rate variability at minutes -25 to -20; Test type: Superiority; p = 0.3139, t-test, 2 sided
Statistical Analysis 5: Comparison: Intranasal Oxytocin vs Placebo; High frequency heart rate variability at minutes -20 to -15; Test type: Superiority; p = 0.4222, t-test, 2 sided
Statistical Analysis 6: Comparison: Intranasal Oxytocin vs Placebo; High frequency heart rate variability at minutes -15 to -10; Test type: Superiority; p = 0.834, t-test, 2 sided
Statistical Analysis 7: Comparison: Intranasal Oxytocin vs Placebo; High frequency heart rate variability at minutes -10 to -5; Test type: Superiority; p = 0.7562, t-test, 2 sided
Statistical Analysis 8: Comparison: Intranasal Oxytocin vs Placebo; High frequency heart rate variability at minutes -5 to 0; Test type: Superiority; p = 0.4245, t-test, 2 sided
Statistical Analysis 9: Comparison: Intranasal Oxytocin vs Placebo; High frequency heart rate variability at minutes 5 to 8; Test type: Superiority; p = 0.1425, t-test, 2 sided
Statistical Analysis 10: Comparison: Intranasal Oxytocin vs Placebo; High frequency heart rate variability at minutes 8 to 13; Test type: Superiority; p = 0.7175, t-test, 2 sided
Statistical Analysis 11: Comparison: Intranasal Oxytocin vs Placebo; High frequency heart rate variability at minutes 13 to 18; Test type: Superiority; p = 0.1417, t-test, 2 sided
Statistical Analysis 12: Comparison: Intranasal Oxytocin vs Placebo; High frequency heart rate variability at minutes 18 to 23; Test type: Superiority; p = 0.0514, t-test, 2 sided
Statistical Analysis 13: Comparison: Intranasal Oxytocin vs Placebo; High frequency heart rate variability at minutes 23 to 28; Test type: Superiority; p = 0.1507, t-test, 2 sided
Statistical Analysis 14: Comparison: Intranasal Oxytocin vs Placebo; High frequency heart rate variability at minutes 8 to 33; Test type: Superiority; p = 0.4204, t-test, 2 sided
Statistical Analysis 15: Comparison: Intranasal Oxytocin vs Placebo; High frequency heart rate variability at minutes 33 to 38; Test type: Superiority; p = 0.4209, t-test, 2 sided
Statistical Analysis 16: Comparison: Intranasal Oxytocin vs Placebo; High frequency heart rate variability at minutes 38 to 43; Test type: Superiority; p = 0.2569, t-test, 2 sided
Statistical Analysis 17: Comparison: Intranasal Oxytocin vs Placebo; High frequency heart rate variability at minutes 43 to 48; Test type: Superiority; p = 0.0828, t-test, 2 sided

5. Secondary Outcome: Changes in Pre-ejection Period, an Index of Sympathetic Activity, During the TSST
Description: Recording of autonomic activity beginning prior to study drug administration (-40 minutes) until the end of recovery from the TSST (+38 minutes). Mobile Impedance Cardiographs (MindWare Tech Ltd, Gahanna, OH) will be used to measure pre-ejection period (PEP). PEP will index sympathetic activation. Results are reported as difference from the mean of pre-ejection period measured in the first ten minutes of the study visit, prior to administration of OT or placebo.
Time Frame: as for outcome 4
Population: For some participants in each arm, cardiograph recording was unsuccessful. For some time periods for some participants, data quality or quantity (in terms of lacking sufficient numbers of epochs within a period) was insufficient for analysis. All valid, analyzable data are reported herein.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Intranasal Oxytocin | Placebo
Number analyzed (Participants) | 46 | 39
milliseconds
  -40 to -35: number analyzed (Participants) | 45 | 39
  -40 to -35 | -0.0133 (5.0895) | -0.5344 (5.2068)
  -35 to -30: number analyzed (Participants) | 44 | 39
  -35 to -30 | -0.4379 (4.6949) | -1.578 (5.6245)
  -30 to -25: number analyzed (Participants) | 44 | 39
  -30 to -25 | -0.0765 (4.8828) | -1.2421 (6.3071)
  -25 to -20: number analyzed (Participants) | 43 | 39
  -25 to -20 | 0.1364 (5.4471) | -0.9139 (6.4616)
  -20 to -15: number analyzed (Participants) | 42 | 39
  -20 to -15 | 0.4913 (6.0127) | -0.743 (5.4354)
  -15 to -10: number analyzed (Participants) | 42 | 37
  -15 to -10 | 0.396 (6.5937) | -1.2658 (6.5275)
  -10 to -5: number analyzed (Participants) | 42 | 38
  -10 to -5 | 0.1857 (5.745) | -1.9649 (6.0961)
  -5 to 0: number analyzed (Participants) | 42 | 37
  -5 to 0 | 0.7484 (5.8793) | -2.3991 (5.8181)
  5 to 8: number analyzed (Participants) | 42 | 36
  5 to 8 | -4.9659 (7.7046) | -6.9426 (14.7706)
  8 to 13: number analyzed (Participants) | 41 | 38
  8 to 13 | -4.9797 (14.7581) | -6.7011 (12.5175)
  13 to 18: number analyzed (Participants) | 41 | 38
  13 to 18 | -4.4699 (14.2813) | -7.2932 (12.2579)
  18 to 23: number analyzed (Participants) | 43 | 38
  18 to 23 | 0.3473 (6.8964) | -1.7225 (5.6289)
  23 to 28: number analyzed (Participants) | 40 | 37
  23 to 28 | 1.0633 (5.9026) | -0.5384 (5.2814)
  28 to 33: number analyzed (Participants) | 40 | 37
  28 to 33 | 1.47 (5.9291) | -0.3492 (4.7881)
  33 to 38: number analyzed (Participants) | 40 | 37
  33 to 38 | 1.1908 (5.6515) | -0.706 (4.7005)
  38 to 43: number analyzed (Participants) | 39 | 37
  38 to 43 | 1.3179 (5.8975) | -0.3979 (4.7213)
  43 to 48: number analyzed (Participants) | 39 | 37
  43 to 48 | 1.2028 (5.8875) | -0.833 (4.2802)
Statistical Analysis 1: Comparison: Intranasal Oxytocin vs Placebo; Pre-ejection period at minutes -40 to -35; Test type: Superiority; p = 0.6452, t-test, 2 sided
Statistical Analysis 2: Comparison: Intranasal Oxytocin vs Placebo; Pre-ejection period at minutes -35 to -30; Test type: Superiority; p = 0.3228, t-test, 2 sided
Statistical Analysis 3: Comparison: Intranasal Oxytocin vs Placebo; Pre-ejection period at minutes -30 to -25; Test type: Superiority; p = 0.3541, t-test, 2 sided
Statistical Analysis 4: Comparison: Intranasal Oxytocin vs Placebo; Pre-ejection period at minutes -25 to -20; Test type: Superiority; p = 0.4311, t-test, 2 sided
Statistical Analysis 5: Comparison: Intranasal Oxytocin vs Placebo; Pre-ejection period at minutes -20 to -15; Test type: Superiority; p = 0.3349, t-test, 2 sided
Statistical Analysis 6: Comparison: Intranasal Oxytocin vs Placebo; Pre-ejection period at minutes -15 to -10; Test type: Superiority; p = 0.2646, t-test, 2 sided
Statistical Analysis 7: Comparison: Intranasal Oxytocin vs Placebo; Pre-ejection period at minutes -10 to -5; Test type: Superiority; p = 0.1095, t-test, 2 sided
Statistical Analysis 8: Comparison: Intranasal Oxytocin vs Placebo; Pre-ejection period at minutes -5 to 0; Test type: Superiority; p = 0.0194, t-test, 2 sided
Statistical Analysis 9: Comparison: Intranasal Oxytocin vs Placebo; Pre-ejection period at minutes 5 to 8; Test type: Superiority; p = 0.473, t-test, 2 sided
Statistical Analysis 10: Comparison: Intranasal Oxytocin vs Placebo; Pre-ejection period at minutes 8 to 13; Test type: Superiority; p = 0.5768, t-test, 2 sided
Statistical Analysis 11: Comparison: Intranasal Oxytocin vs Placebo; Pre-ejection period at minutes 13 to 18; Test type: Superiority; p = 0.3477, t-test, 2 sided
Statistical Analysis 12: Comparison: Intranasal Oxytocin vs Placebo; Pre-ejection period at minutes 18 to 23; Test type: Superiority; p = 0.1413, t-test, 2 sided
Statistical Analysis 13: Comparison: Intranasal Oxytocin vs Placebo; Pre-ejection period at minutes 23 to 28; Test type: Superiority; p = 0.2128, t-test, 2 sided
Statistical Analysis 14: Comparison: Intranasal Oxytocin vs Placebo; Pre-ejection period at minutes 28 to 33; Test type: Superiority; p = 0.1415, t-test, 2 sided
Statistical Analysis 15: Comparison: Intranasal Oxytocin vs Placebo; Pre-ejection period at minutes 33 to 38; Test type: Superiority; p = 0.1126, t-test, 2 sided
Statistical Analysis 16: Comparison: Intranasal Oxytocin vs Placebo; Pre-ejection period at minutes 38 to 43; Test type: Superiority; p = 0.1647, t-test, 2 sided
Statistical Analysis 17: Comparison: Intranasal Oxytocin vs Placebo; Pre-ejection period at minutes 43 to 48; Test type: Superiority; p = 0.088, t-test, 2 sided

6. Other Pre Specified Outcome: Assessment of Effect Modification by Maternal Depression / Anxiety on Changes in Cortisol (CRT) During Trier Social Stress Test (TSST)
Description: Stratified analyses will be performed to determine the extent to which maternal depression/anxiety modifies the effect of OT/placebo on CRT during the TSST.
Time Frame: -40 minutes, -20 minutes, 0 minutes, +10 minutes, +15 minutes, +28 minutes, +38 minutes, +48 minutes
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Assessment of Effect Modification by Maternal Depression / Anxiety on Changes in Adrenocorticotropic Hormone (ACTH ) During TSST
Description: Stratified analyses will be performed to determine the extent to which maternal depression/anxiety modifies the effect of OT/placebo on ACTH during the TSST.
Time Frame: -40 minutes, -20 minutes, 0 minutes, +10 minutes, +15 minutes, +28 minutes, +38 minutes, +48 minutes
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Assessment of Effect Modification by Maternal Depression / Anxiety on Changes in High Frequency Heart Rate Variability, an Index of Parasympathetic Activity, During the TSST
Description: Stratified analyses will be performed to determine the extent to which maternal depression/anxiety modifies the effect of OT/placebo on parasympathetic activity during the TSST.
Time Frame: Minutes -40 to -35, -35 to -30, -30 to -25, -25 to -20, -20 to -15, -15 to -10, -10 to -5, -5 to 0, 0 to 5, 5 to 8, 8 to 13, 13 to 18, 18 to 23, 23 to 28, 28 to 33, 33 to 38, 38 to 43, 43 to 48
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Assessment of Effect Modification by Maternal Depression / Anxiety on Changes in Pre-ejection Period, an Index of Sympathetic Activity, During the TSST
Description: Stratified analyses will be performed to determine the extent to which maternal depression/anxiety modifies the effect of OT/placebo on sympathetic activity during the TSST.
Time Frame: as for outcome 8
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Assessment of Effect Modification by Oxytocin Receptor (OXTR) Genotype on Changes in Cortisol (CRT) During Trier Social Stress Test (TSST)
Description: as for outcome 6
Time Frame: -40 minutes, -20 minutes, 0 minutes, +10 minutes, +15 minutes, +28 minutes, +38 minutes, +48 minutes
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Assessment of Effect Modification by OXTR Genotype on Changes in Adrenocorticotropic Hormone (ACTH ) During TSST
Description: as for outcome 7
Time Frame: -30 minutes, 0 minutes, +10 minutes, +15 minutes, +28 minutes, +38 minutes
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Assessment of Effect Modification by OXTR Genotype Changes in High Frequency Heart Rate Variability, an Index of Parasympathetic Activity, During the TSST
Description: as for outcome 8
Time Frame: as for outcome 8
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Assessment of Effect Modification by OXTR Genotype on Changes in Pre-ejection Period, an Index of Sympathetic Activity, During the TSST
Description: as for outcome 9
Time Frame: as for outcome 8
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From the time of study drug administration through the end of the recovery period, a total of approximately 90 minutes.
Arm/Group | Intranasal Oxytocin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/54
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/54
Other Adverse Events (participants affected / at risk) | 0/51 | 1/54
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intranasal Oxytocin (N=51) | Placebo (N=54)
Hypotension (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-01-19): https://cdn.clinicaltrials.gov/large-docs/73/NCT03593473/Prot_SAP_001.pdf
  • Informed Consent Form (2022-12-08): https://cdn.clinicaltrials.gov/large-docs/73/NCT03593473/ICF_000.pdf